CLINICAL TRIAL: NCT00516776
Title: The Innate Immune System and Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 5.2007.910
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Intestinal biopsies Plasma/serum Peripheral blood monocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study includes individuals with ulcerative colitis, Crohn's disease and healthy controls. The purpose of this study is to examine the innate immune system (IIS) by exposing peripheral blood monocytes to various ligands relevant for stimulation of the IIS and study the immune response. Colonic mucosal samples are examined to find gene expression patterns which may distinguish the two forms of disease from each other and from healthy controls.

The hypothesis is that the innate immune system has responses unique for the disease states, and that the diseases may be differentiated by examination of gene expression patterns in mucosal biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ulcerative colitis
* Presence of Crohn's disease
* Healthy (no sign of inflammatory bowel disease)

Exclusion Criteria:

* Anticoagulation
* Cardiac valvular disease
* Intravascular prosthesis
* Coagulation disorders
* Gastrointestinal malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from endoscopy unit and outpatients clinic with ulcerative colitis, Crohn's disease and healthy controls
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
gene expression patterns in mucosal biopsies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arne K Sandvik, MD PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Dept of Cancer Research and Molecular Medicine, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brenna O, Bruland T, Furnes MW, Granlund Av, Drozdov I, Emgard J, Bronstad G, Kidd M, Sandvik AK, Gustafsson BI. The guanylate cyclase-C signaling pathway is down-regulated in inflammatory bowel disease. Scand J Gastroenterol. 2015;50(10):1241-52. doi: 10.3109/00365521.2015.1038849. Epub 2015 May 15. PMID 25979109
- [Derived] Ostvik AE, Granlund Av, Gustafsson BI, Torp SH, Espevik T, Mollnes TE, Damas JK, Sandvik AK. Mucosal toll-like receptor 3-dependent synthesis of complement factor B and systemic complement activation in inflammatory bowel disease. Inflamm Bowel Dis. 2014 Jun;20(6):995-1003. doi: 10.1097/MIB.0000000000000035. PMID 24739633
- [Derived] Ostvik AE, Granlund AV, Bugge M, Nilsen NJ, Torp SH, Waldum HL, Damas JK, Espevik T, Sandvik AK. Enhanced expression of CXCL10 in inflammatory bowel disease: potential role of mucosal Toll-like receptor 3 stimulation. Inflamm Bowel Dis. 2013 Feb;19(2):265-74. doi: 10.1002/ibd.23034. PMID 22685032